CLINICAL TRIAL: NCT05085236
Title: Therapeutic Effect of Fu's Subcutaneous Needling for Recovery Outcomes of Stroke Survivors With Hemiplegic Shoulder Pain.: Randomized-controlled Trial
Brief Title: Fu's Subcutaneous Needling Treatment for Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC2-124
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-08

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Fu's subcutaneous needling; post-stroke complications; post-stroke shoulder pain; hemiplegic shoulder pain; shoulder hand syndrome
MeSH Terms: conditions — Reflex Sympathetic Dystrophy | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu's subcutaneous needling (FSN) in combination with rehabilitation (Experimental): In this arm, the subjects will receive the intervention of FSN combined with regular rehabilitation program on Day1, Day2, and Day4, in total 3 treatments. The subjects will receive assessments before and after each interventions. After total treatments finishing, the subjects will receive assessments on Day8 and Day15.
  Interventions: Procedure: Fu's subcutaneous needling (FSN); Procedure: Rehabilitation
- Rehabilitation (Active Comparator): In this arm, the subjects will receive the intervention of regular rehabilitation program prescribed by physician of rehabilitation. On Day1, Day2, and Day4, the subjects will receive assessments before and after each interventions. After total treatments finishing, the subjects will receive assessments on Day8 and Day15.
  Interventions: Procedure: Rehabilitation

INTERVENTIONS:
Procedure: Fu's subcutaneous needling (FSN) — physician will use a disposable Fu's subcutaneous needling (FSN) to penetrate the subject's skin in the middle from elbow lateral epicondyle to radial styloid process. Then physician will push forward the needle parallel to the skin surface. the physician will sway the needle 100 times in a minute. After procedure of swaying needle, the physician will instruct subject to do several movements, and each movement will perform 10 seconds and rest 10 seconds for 3 repetitions. The movements are active isometric elbow flexion, active isometric shoulder internal rotation, passive shoulder external and internal rotation. After above re-perfusion approach of muscles, the physician will take out the needle to finish the treatment.
  Arms: Fu's subcutaneous needling (FSN) in combination with rehabilitation
Procedure: Rehabilitation — Rehabilitation mentioned here is the regular rehabilitation programs for treating post-stroke hemiplegic shoulder pain prescribed by the rehabilitation physician.

SUMMARY:
The post-stroke survivors suffered from shoulder pain are very common. The investigators performed Fu's subcutaneous needling (FSN). This experiment used a randomized controlled trial to assess the immediate, short-term and long-term effects of Fu's subcutaneous needling therapy on hemiplegic shoulder pain in patient with stroke.

DETAILED DESCRIPTION:
The prevalence of complication in post-stroke survivors is 30-96%. Post-stroke pain is the most common complication. According to previous researches there are sixty percent post-stroke survivors who suffered from upper limb pain. The mechanism causes post-stroke shoulder pain is imbalance of shoulder muscles and in-coordination of shoulder motor control due to cerebral vascular disease. Post-stroke shoulder pain often causes the limitation of shoulder range of motion, and the pain always affected quality of life and daily activities. Because of shoulder pain, those post-stroke survivors postponed the program of rehabilitation. The treatments of post-stroke shoulder pain are transcutaneous electrical nerve stimulation, drug, intra-articular injection and nerve block. Acupuncture with combination of rehabilitation has been proved by many researches in alleviating pain and increasing quality of life in treating post-stroke shoulder pain. Fu's subcutaneous needling is a newly technique based on meridian theory and the technique is used to treat cervical, lumbar and four limb's pain proved by many researches. Fu's subcutaneous needling in managing post-stroke pain has less reported, so investigator set up a proposal to see if the Fu's subcutaneous needling could elevate more therapeutic effect compared to usual care or not.

The investigators will enroll patients into two groups, experimental and control groups. The interventions in experimental group are Fu's subcutaneous needling in combination with rehabilitation, and in control group is rehabilitation. The trial will extend two weeks, and investigator will treat with Fu's subcutaneous needling three times in the first, second and fourth day when the patients include to our trial. The outcome measurements are visual analog scale, range of motion of shoulder, pressure pain threshold of myofascial trigger point, acromion-greater tuberosity distance, Fugl-Meyer assessment in upper extremity and functional independence measure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteers who are older than 40 years old suffered from first stroke attack including infarction and hemorrhage with image proved and can cooperate with the experiment.
* 2. Stroke patient suffered from shoulder pain.
* 3. Patient can follow the directions of Fu's subcutaneous needling and regular rehabilitation program.

Exclusion Criteria:

* 1. There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant and lactated women.
* 2. There has been a history of drug abuse (including excess alcohol) that affects pain assessment.
* 3. Cognitive impairment, unable to cooperate with the experiment.
* 4. Aphasia
* 5. Have received shoulder joint injection in recent 6 months.
* 6. Have serious skin infection, laceration, wound and trauma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 day
  A Visual Analog Scale consists of a line, often 10 cm long, with verbal anchors at either end, on left of line, zero, meant no pain otherwise on right, 10, meant strong pain. The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Pressure Pain Threshold | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom
Range of Motion of Shoulder | 1 day
  Range of Motion is the measurement of movement around a specific joint, measured in degrees of a circle. In this study we measure shoulder joint, glenohumeral joint, in flexion, extension, external and internal rotation.
Acromion-GreaterTuberosity Distance | 1 day
  In this study we assess of shoulder joint subluxation by means of ultrasound measurement of Acromion-greater tuberosity distance.
Fugl-Meyer assessment in upper extremity | 1 day
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. In upper extremity, we measure motor function included shoulder, elbow, wrist and hand, and assess coordination using finger to nose.
Functional Independence Measure | 1 day
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability. Includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided